CLINICAL TRIAL: NCT05534321
Title: Prophylactic Radiotherapy of MInimally Symptomatic Spinal Disease (PROMISSeD Trial)
Brief Title: Prophylactic Radiotherapy of MInimally Symptomatic Spinal Disease
Acronym: PROMISSeD
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Baptist Health South Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2021-KOT-002
Record Dates: First submitted 2022-09-06; First posted 2022-09-09 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-01

CONDITIONS: Spine Metastases
Keywords: Radiotherapy (RT); Palliative radiotherapy; High-risk asymptomatic spine metastases; Minimal asymptomatic spine metastases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Standard of Care Systemic Therapy or Surveillance (Active Comparator): Patients randomized to arm 1 will undergo appropriate systemic therapy as determined by their oncology team. These patients will either continue the current therapy or be transitioned to a new standard of care therapy at the discretion of the treating oncologist. If randomized to arm 1, these patients may also undergo palliative radiation therapy for progressive or painful lesions (a skeletal related event as defined in the study) at the time of symptom development*(not upfront palliative radiation therapy)
  Interventions: Drug: Standard of care systemic therapy
- Prophylactic Radiation Therapy (Experimental): Patients randomized to Arm 2 of the study will undergo upfront prophylactic radiotherapy to ≤ 5 highest risk bone metastases followed by standard of care, as defined by:
  1. Bulkiest sites of disease ≥ 2cm (can include paraspinal disease extension)
  2. Disease in junctional spine (Occ-C2, C7-T1, T12-L1, L5-S1)
  3. Disease with posterior element involvement (facet(s), interspinous)
  4. Compression Deformity > 50%
  Interventions: Radiation: Prophylactic Radiotherapy

INTERVENTIONS:
Radiation: Prophylactic Radiotherapy — Radiation therapy will be delivered according to department standards. For this protocol, total dose and dose fractionation may be delivered at the discretion of the treating radiation oncologist according to department standards. All techniques including conventional, three-dimensional conformal radiation therapy (3D-CRT), intensity-modulated radiation therapy (IMRT), and stereotactic radiosurgery/stereotactic body radiation therapy (SRS/SBRT) techniques may be used. Image guidance at the time of treatment delivery to verify patient positioning may be chosen at the discretion of the treating radiation oncologist according to department standards.
  Arms: Prophylactic Radiation Therapy
Drug: Standard of care systemic therapy — Standard of care systemic therapy, including chemotherapeutics, targeted therapies, immunomodulatory agents, and hormonal therapies will be delivered at the discretion of the treating medical oncologist. Patients may receive systemic therapy concurrently and there are no restrictions on initiation of systemic agents after radiotherapy including immunotherapy and hormonal therapy, the timing of which will be determined by a consensus between the treating medical and radiation oncologists.
  Arms: Standard of Care Systemic Therapy or Surveillance

SUMMARY:
Early palliative care has been shown to improve the quality of life and even survival for patients with metastatic cancer. More and more supportive oncology teams in cancer centers now advocate for early integration of radiation therapy (RT) in a patient's palliative management course. While multiple randomized studies have evaluated the efficacy of different RT regimens in the treatment of symptomatic bone lesions, few studies have examined the impact of early, upfront RT for asymptomatic or minimally symptomatic (non- opioid dependent) spine metastases and its efficacy in preventing skeletal-related events (SREs). Since the pathophysiology of spinal metastatic disease is distinct from other bony metastatic disease, the proposed trial seeks to understand whether it is beneficial to patients with minimally symptomatic disease to undergo upfront RT to reduce the risks of SREs and their sequelae, including hospitalizations.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically-confirmed solid tumor malignancy with greater than 5 sites of metastatic disease detected on cross-sectional imaging.
2. Has high-risk bone metastases that are asymptomatic or minimally symptomatic (not requiring opioids). High risk metastases are defined as:

   1. Bulkiest sites of spinal osseous disease ≥ 2cm,
   2. Disease at junctional levels, including the thoracic apex (Occiput to C2, C7-T1, T12-L2, and L5- S1)
   3. Disease with posterior element involvement, including interspinous, unilateral, or bilateral facet joints.
   4. Vertebral body compression deformity > 50%.
3. Eastern Cooperative Oncology Group (ECOG) performance status 0 - 2.
4. Age ≥ 18 years.
5. Able to provide informed consent.
6. Patients at reproductive potential must agree to practice an effective contraceptive method. Women of childbearing potential must not be pregnant or lactating.

Exclusion Criteria:

1. Previous RT to the intended treatment site that precludes developing a treatment plan that respects normal tissue tolerances.
2. Serious medical co-morbidities precluding RT.
3. Pregnant or lactating women.
4. Target lesion(s) is/are complicated bone metastases that include clinical or radiological evidence of spinal cord compression or impending pathological fracture.
5. Leptomeningeal disease.
6. Patients whose entry to the trial will cause unacceptable clinical delays in their planned management.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2022-08-29 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Number of patients who have skeletal-related events (SREs) | 1 year
  Number of skeletal related events (SREs), which will be defined as pathological fractures, spinal cord compression, or interventions (palliative RT, interventional procedures, or spine surgery)

SECONDARY OUTCOMES:
Number of skeletal-related event (SRE) hospitalizations | 1 year
  Number of hospitalizations attributed to skeletal-related events (SREs)
Pain-related quality of life | 3 months, 6 months, and 12 months, optionally within 1 week of a skeletal-related event (SRE)
  Pain-related quality of life using the Brief Pain Inventory (BPI) form. The BPI is a 17-item patient self-rating scale assessing demographic data, use of medications, as well as the sensory and reactive components of pain. The scale is from 0-10, and there are breakpoints between scores of 4 and 5 and between 6 and 7, indicating that mild pain correlates with scores of 1-4, moderate pain with 5-6, and severe pain with scores of 7-10.
Health care utilities and quality of life | 3 months, 6 months, and 12 months, optionally within 1 week of a skeletal-related event (SRE)
  Health care utilities and quality of life using the EuroQol Group EQ-5D-5L form. It has been developed to generate a generic cardinal index of health, thus giving it considerable potential for future use in economic evaluation. The EQ-5D-5L is a two-part, patient-completed questionnaire. The first part consists of 5 items covering 5 dimensions including: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension can be graded on 3 levels including: 1=no problems; 2= moderate problems; and 3=extreme problems. The second component is the visual analog scale, where the participant rates their own overall health on a scale of 0 (worst health) to 100 (best health).
Pain-free survival (PFS) | Until 1 year
  Pain-free survival (PFS) is defined as the time from study entry to until the start of opioid use or until death.
Overall survival (OS) | Until 1 year
  Overall survival (OS) is defined as the time from study entry until death.
Adverse event frequency and severity | 3 months, 6 months, and 12 months
  Evaluate CTCAE v5 toxicity events in the upfront RT arm by tabulating all toxicities and summarizing the CTCAE v5 scores.

CONTACTS AND LOCATIONS:
Overall Officials: Rupesh R Kotecha, MD, Principal Investigator — Miami Cancer Institute
Locations (1):
- Miami Cancer Institute at Baptist Health South Florida, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Mundy GR. Metastasis to bone: causes, consequences and therapeutic opportunities. Nat Rev Cancer. 2002 Aug;2(8):584-93. doi: 10.1038/nrc867. PMID 12154351
- [Background] Lutz ST, Jones J, Chow E. Role of radiation therapy in palliative care of the patient with cancer. J Clin Oncol. 2014 Sep 10;32(26):2913-9. doi: 10.1200/JCO.2014.55.1143. Epub 2014 Aug 11. PMID 25113773
- [Background] Lutz S, Balboni T, Jones J, Lo S, Petit J, Rich SE, Wong R, Hahn C. Palliative radiation therapy for bone metastases: Update of an ASTRO Evidence-Based Guideline. Pract Radiat Oncol. 2017 Jan-Feb;7(1):4-12. doi: 10.1016/j.prro.2016.08.001. Epub 2016 Aug 5. PMID 27663933
- [Background] Rades D, Segedin B, Conde-Moreno AJ, Garcia R, Perpar A, Metz M, Badakhshi H, Schreiber A, Nitsche M, Hipp P, Schulze W, Adamietz IA, Norkus D, Rudat V, Cacicedo J, Schild SE. Radiotherapy With 4 Gy x 5 Versus 3 Gy x 10 for Metastatic Epidural Spinal Cord Compression: Final Results of the SCORE-2 Trial (ARO 2009/01). J Clin Oncol. 2016 Feb 20;34(6):597-602. doi: 10.1200/JCO.2015.64.0862. Epub 2016 Jan 4. PMID 26729431
- [Background] Zimmermann C, Swami N, Krzyzanowska M, Hannon B, Leighl N, Oza A, Moore M, Rydall A, Rodin G, Tannock I, Donner A, Lo C. Early palliative care for patients with advanced cancer: a cluster-randomised controlled trial. Lancet. 2014 May 17;383(9930):1721-30. doi: 10.1016/S0140-6736(13)62416-2. Epub 2014 Feb 19. PMID 24559581
- [Background] Rothrock RJ, Reiner AS, Barzilai O, Kim NC, Ogilvie SQ, Lis E, Gulati A, Yamada Y, Bilsky MH, Laufer I. Responder Analysis of Pain Relief After Surgery for the Treatment of Spinal Metastatic Tumors. Neurosurgery. 2022 Oct 1;91(4):604-617. doi: 10.1227/neu.0000000000002083. Epub 2022 Jul 22. PMID 35856981
- [Background] Lipton A, Theriault RL, Hortobagyi GN, Simeone J, Knight RD, Mellars K, Reitsma DJ, Heffernan M, Seaman JJ. Pamidronate prevents skeletal complications and is effective palliative treatment in women with breast carcinoma and osteolytic bone metastases: long term follow-up of two randomized, placebo-controlled trials. Cancer. 2000 Mar 1;88(5):1082-90. doi: 10.1002/(sici)1097-0142(20000301)88:53.0.co;2-z. PMID 10699899
- [Background] Saad F, Gleason DM, Murray R, Tchekmedyian S, Venner P, Lacombe L, Chin JL, Vinholes JJ, Goas JA, Zheng M; Zoledronic Acid Prostate Cancer Study Group. Long-term efficacy of zoledronic acid for the prevention of skeletal complications in patients with metastatic hormone-refractory prostate cancer. J Natl Cancer Inst. 2004 Jun 2;96(11):879-82. doi: 10.1093/jnci/djh141. PMID 15173273
- [Background] Rosen LS, Gordon D, Tchekmedyian NS, Yanagihara R, Hirsh V, Krzakowski M, Pawlicki M, De Souza P, Zheng M, Urbanowitz G, Reitsma D, Seaman J. Long-term efficacy and safety of zoledronic acid in the treatment of skeletal metastases in patients with nonsmall cell lung carcinoma and other solid tumors: a randomized, Phase III, double-blind, placebo-controlled trial. Cancer. 2004 Jun 15;100(12):2613-21. doi: 10.1002/cncr.20308. PMID 15197804
- [Background] Saad F, Lipton A. Zoledronic acid is effective in preventing and delaying skeletal events in patients with bone metastases secondary to genitourinary cancers. BJU Int. 2005 Nov;96(7):964-9. doi: 10.1111/j.1464-410X.2005.05740.x. PMID 16225510
- [Background] Duran I, Fink MG, Bahl A, Hoefeler H, Mahmood A, Luftner D, Ghazal H, Wei R, Chung KC, Hechmati G, Green J, Atchison C. Health resource utilisation associated with skeletal-related events in patients with bone metastases secondary to solid tumours: regional comparisons in an observational study. Eur J Cancer Care (Engl). 2017 Nov;26(6). doi: 10.1111/ecc.12452. Epub 2016 Feb 10. PMID 26865392
- [Background] Luftner D, Lorusso V, Duran I, Hechmati G, Garzon-Rodriguez C, Ashcroft J, Bahl A, Ghelani P, Wei R, Thomas E, Hoefeler H. Health resource utilization associated with skeletal-related events in patients with advanced breast cancer: results from a prospective, multinational observational study. Springerplus. 2014 Jun 30;3:328. doi: 10.1186/2193-1801-3-328. eCollection 2014. PMID 25045611
- [Background] Stopeck A, Rader M, Henry D, Danese M, Halperin M, Cong Z, Qian Y, Dansey R, Chung K. Cost-effectiveness of denosumab vs zoledronic acid for prevention of skeletal-related events in patients with solid tumors and bone metastases in the United States. J Med Econ. 2012;15(4):712-23. doi: 10.3111/13696998.2012.675380. Epub 2012 Mar 27. PMID 22409231
- [Background] Degen JW, Gagnon GJ, Voyadzis JM, McRae DA, Lunsden M, Dieterich S, Molzahn I, Henderson FC. CyberKnife stereotactic radiosurgical treatment of spinal tumors for pain control and quality of life. J Neurosurg Spine. 2005 May;2(5):540-9. doi: 10.3171/spi.2005.2.5.0540. PMID 15945428
- [Background] Daut RL, Cleeland CS, Flanery RC. Development of the Wisconsin Brief Pain Questionnaire to assess pain in cancer and other diseases. Pain. 1983 Oct;17(2):197-210. doi: 10.1016/0304-3959(83)90143-4. PMID 6646795
- [Background] Jensen MP, Turner JA, Romano JM, Fisher LD. Comparative reliability and validity of chronic pain intensity measures. Pain. 1999 Nov;83(2):157-62. doi: 10.1016/s0304-3959(99)00101-3. PMID 10534586
- [Background] Cleeland CS. Measurement of pain by subjective report. In: Chapman CR; Loeser JD, editors. Issues in pain measurement. New York: Raven Press; 1989: 391-403.
- [Background] Cella DF, Tulsky DS, Gray G, Sarafian B, Linn E, Bonomi A, Silberman M, Yellen SB, Winicour P, Brannon J, et al. The Functional Assessment of Cancer Therapy scale: development and validation of the general measure. J Clin Oncol. 1993 Mar;11(3):570-9. doi: 10.1200/JCO.1993.11.3.570. PMID 8445433
- [Background] Rabin R, de Charro F. EQ-5D: a measure of health status from the EuroQol Group. Ann Med. 2001 Jul;33(5):337-43. doi: 10.3109/07853890109002087. PMID 11491192
- [Background] Badia X, Herdman M, Kind P. The influence of ill-health experience on the valuation of health. Pharmacoeconomics. 1998 Jun;13(6):687-96. doi: 10.2165/00019053-199813060-00005. PMID 10179704
- [Background] Mirels H. Metastatic disease in long bones. A proposed scoring system for diagnosing impending pathologic fractures. Clin Orthop Relat Res. 1989 Dec;(249):256-64. PMID 2684463
- [Derived] Rothrock RJ, Ozair A, Avendano MC, Herrera S, Appel H, Ramos S, Starosciak AK, Leon-Ariza DS, Rubens M, McDermott MW, Ahluwalia MS, Mehta MP, Kotecha RR. Prophylactic Radiotherapy Of MInimally Symptomatic Spinal Disease (PROMISSeD): study protocol for a randomized controlled trial. Trials. 2024 Jan 12;25(1):41. doi: 10.1186/s13063-023-07850-8. PMID 38217032